CLINICAL TRIAL: NCT04105478
Title: Early Migration of Stemless and Stemmed Humeral Components After Total Shoulder Arthroplasty for Osteoarthritis - A Randomized Controlled Trial
Brief Title: Comparison of Stemless and Stemmed Shoulder Arthroplasty for Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Marc Randall Kristensen Nyring, Principal investigator, PhD student, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nano study
Record Dates: First submitted 2019-09-17; First posted 2019-09-26 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Glenohumeral Osteoarthritis
MeSH Terms: interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Intervention Model Description: Based on the sample calculation the investigators intend to include a total number of 122 patients of which the first 56 patients will be studied using MB-RSA and DXA. The patients are allocated into two groups of equal of size:
  1. The un-cemented Comprehensive Nano stemless shoulder arthroplasty (intervention group)
  2. The un-cemented Comprehensive stemmed total shoulder arthroplasty (control group)
  The randomization is done in the operating theater just after the perioperative evaluation of the bone-stock and the rotator cuff. The randomization sequence will be computer generated. The patients will be randomized using stratified, block randomization.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Un-cemented Comprehensive Nano stemless shoulder arthroplasty (Experimental): By using a stemless humeral component stem-related complications can be reduced. Furthermore, the canal preserving design may also facilitate further surgery should the need of a revision prosthesis arise.
  Currently, little is known about the results of the stemless design. The initial results have been promising, but as with the stemmed design migration and eventually loosening of the prosthesis can lead to poor results and, in some cases, revision
  Interventions: Procedure: Shoulder arthroplasty
- Un-cemented Comprehensive stemmed total shoulder arthroplasty (Active Comparator): A design with a metal stem in the humeral bone canal is currently regarded as the best treatment option, but complications related to the stem including humeral fractures can have devastating consequences.
  Interventions: Procedure: Shoulder arthroplasty

INTERVENTIONS:
Procedure: Shoulder arthroplasty — Patients suffering from severe glenohumeral osteoarthritis are treated surgically by a total shoulder arthroplasty

SUMMARY:
This is a randomized controlled trial comparing the Comprehensive Nano stemless total shoulder arthroplasty (intervention group) with the Comprehensive un-cemented stemmed total shoulder arthroplasty (control group). All Danish citizens with glenohumeral osteoarthritis indicating a total shoulder arthroplasty referred to the orthopedic department at Copenhagen University Hospital in Gentofte will be offered participation in the trial. The following exclude from participation in the study: below 18 years of age; cognitive or linguistic impairment; insufficient function of the rotator cuff; poor bone quality and ASA group 4-5. A total of 122 patients will be included of which 56 will be part of radiostereometric analysis (RSA) study of humeral component migration. This will allow a maximum of 20% drop out. The primary outcome is magnitude and pattern of migration of the humeral component assessed by RSA. The secondary outcomes are patient-reported outcomes, functional outcome, readmission, complications, revisions, changes in bone mineral density (BMD) of the proximal humerus assessed by duel energy x-ray absorptiometry (DXA) and economy (cost utility analysis). To avoid bias in some of these outcomes, the patient will not know what type of humeral component was used. The patients are examined before the operation and 3, 6, 12 and 24 months after the operation.

DETAILED DESCRIPTION:
Background Osteoarthritis (wear and tear) of the shoulder can, in the most severe cases, require insertion of shoulder prosthesis (an artificial shoulder joint, a total shoulder arthroplasty). This is an effective treatment with pain-relief and significant improvement in shoulder function. A design with a metal stem in the humeral bone canal is currently regarded as the best treatment option, but complications related to the stem including humeral fractures can have devastating consequences. By using a stemless humeral component stem-related complications can be reduced. Furthermore, the canal preserving design may also facilitate further surgery should the need of a revision prosthesis arise.

Currently, little is known about the results of the stemless design. The initial results have been promising, but as with the stemmed design migration and eventually loosening of the prosthesis can lead to poor results and, in some cases, revision.

Using radiostereometric analysis (RSA) a special x-ray examination technique based upon insertion of small metal beads into the bone surrounding an implant and attachment of beads to the prosthesis (or using 3-dimensional models of the implant (CAD models) = model-based RSA (MB-RSA)), implant migration can be measured extremely accurate. The RSA technique has previously been used to study migration and loosening of hip and knee prostheses. It has been suggested that RSA should be used to monitor small series of new prostheses the first two years after surgery as a part of a safe phased introduction.

RSA has never been used to access migration of a stemmed or a stemless humeral component nor has the stemmed and the stemless humeral component been compared with regard to pain relief and shoulder function.

Purpose The purpose is to compare the Comprehensive Nano stemless total shoulder prosthesis (intervention group) with the Comprehensive stemmed total shoulder prosthesis (control group).

Method All Danish citizens with shoulder osteoarthritis indicating a total shoulder arthroplasty referred to the orthopedic department at Copenhagen University Hospital in Gentofte will be offered participation in the trial. The following exclude from participation in the study: below 18 years of age, cognitive or linguistic impairment, insufficient function of the rotator cuff (muscles which stabilize the shoulder joint) and severe co-morbidity (ASA-score 4-5).

A total of 122 patients will be included of which 56 will be part of the RSA analysis. This will allow a maximum of 20% drop out. The study will be conducted as a randomized clinical trial (RCT) where each participant by lot will be allocated to one of the two designs. Patients will subsequently be carefully monitored to determine whether there is a difference. The primary outcome is magnitude and pattern of migration of the humeral component assessed by MB-RSA. The secondary outcomes are pain relief, questionnaires (patient-reported outcome), range of movement and strength (functional outcome), readmission, complications, revisions, changes in bone density round the shoulder assessed by duel energy x-ray absorptiometry (DXA) and economy (cost utility analysis). To avoid bias in some of these outcomes, the patient will not know what type of prosthesis was used. The patients are examined before the operation and 3, 6, 12 and 24 months after the operation. The investigators expect short-term publications of early results at about 2 years after inclusion of the last patient.

Ethical considerations Apart from the differences in design, the two groups are treated alike. Today, the two designs are considered equal in the treatment of osteoarthritis. With this study, all patients are at risk of being treated with a prosthesis that subsequent analyses will deem inferior. This is implicit in the study design and there is nothing a priori to suggest which prosthesis is the better.

The standard treatment at the orthopedic department at Copenhagen University Hospital in Gentofte includes preoperative planning with plain radiographs, CT and MRI scans of the glenohumeral joint and follow-up examinations with plain radiographs postoperatively and at 3 months. In addition to this standard treatment the participating patients will have additional radiographic examinations including:

RSA examination at 1 week, 3 months, 6 months, and at 1 and 2 years: 0.04 mSv Plain radiographs at 1 and 2 years: 0.02 mSv DXA scans preoperatively, at 1 week, 3 months, 6 months, and at 1 and 2 years: 0.04 mSv

The background radiation in Denmark is 3 mSv each year. The extra radiation dosage of 0.10 mSv from this study corresponds to the background radiation during approximately 12 days.

The standard treatment at the orthopedic department at Copenhagen University Hospital in Gentofte includes a follow-up examination at 3 months. The participating patients will have additional follow-up examinations at 1 week, 6 months, and at 1 and 2 years. Besides being time consuming this may maintain the patients in a role of being ill. However, the patients will also have the advantage of feeling secure and any uncertainty or problems can be addressed more easily.

The results of the study should be of benefit to future patients with osteoarthritis of the shoulder and thereby also for the use of resources in healthcare. Neither the coordinating investigator nor participating investigators or surgeons have personal economic interests in the study results.

ELIGIBILITY:
Inclusion Criteria:

* All Danish citizens with glenohumeral osteoarthritis indicating a total shoulder arthroplasty referred to the orthopedic department at Copenhagen University Hospital in Gentofte

Exclusion Criteria:

* below 18 years of age
* cognitive or linguistic impairment
* insufficient function of the rotator cuff
* poor bone quality
* ASA group 4-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Radiostereometric analysis (RSA) | Change from 1 week postoperatively to 3 months, 6 months, and at 1 and 2 years postoperatively
  A special x-ray examination technique based upon insertion of small metal beads into the bone surrounding an implant and attachment of beads to the prosthesis (or using 3-dimensional models of the implant (CAD models) = model-based RSA (MB-RSA)). In this way, implant migration can be measured extremely accurate.
Western Ontario Osteoarthritis of the Shoulder index (WOOS) | Change in WOOS score from preoperatively to 3 months, 6 months, and at 1 and 2 years postoperatively
  The WOOS is a disease-specific patient-reported outcome (Lo IK et al 2001). There are 19 questions divided into four domains: Physical symptoms, sports and work, lifestyle and emotions. Each question is answered on a visual analogue scale ranging from 0 to 100. The overall score ranges from 0 to 1900, with 1900 being the worst. For ease of interpretation, the scores are converted to a percentage of the maximum score. We use a Danish version of WOOS (Rasmussen JV et al 2013) which was translated according to the guidelines of Guillemin, Bombardier and Beaton (Guillemin F et al 1993). It was validated with classical test theory in a cohort of patients treated with shoulder arthroplasty for osteoarthritis.

SECONDARY OUTCOMES:
Duel energy x-ray absorptiometry (DXA) | Preoperatively and at 1 week, 3 months, 6 months, and at 1 and 2 years postoperatively
  Changes in bone mineral density (BMD) in close relation to an orthopedic implant can be measured by duel x-ray absorptiometry (DXA)
Plain radiographs | Preoperatively and at 1 week, 3 months and at 1 and 2 years postoperatively
  We use an anterior-posterior and a lateral view. The radiographs are used to evaluate the position of the component and to evaluate loosening as the cause of failure.
Oxford Shoulder Score (OSS) | Preoperatively and 3 months, 6 months, and at 1 and 2 years postoperatively
  Oxford Shoulder Score (OSS): The OSS was conceived as a measurement tool for the assessment of pain and function after elective shoulder surgery (Dawson J et al 1996). There are 12 questions with each item scored from 1-5. The overall score ranges from 12 to 60, with 60 being the worst. For ease of interpretation, the scores are converted to a percentage of the maximum score. We use a Danish version of OSS which was translated and validated with classical test theory (Frich LH et al 2011).
Constant-Murley score | Preoperatively and 3 months, 6 months, and at 1 and 2 years postoperatively
  The Constant-Murley Score includes an assessment of: pain; activities of daily living (ADL); range of motion; and strength. There are a possible 35 points given for the subjective assessment of pain and the ability to perform ADL. There are a possible 65 points given for an objective assessment, of which 40 points are allocated to range of motion and 25 points are allocated to strength. The maximum of 100 point indicates a shoulder with no disability. We use a Danish version (Ban I et al 2013) of the modified score described by Con¬stant and colleagues in 2008 (Constant CR et al 2008).
Pain and patient-satisfaction: visual analogue scale (VAS) | 3 months, 6 months, and at 1 and 2 years postoperatively
  Pain is answered on a visual analogue scale (VAS) ranging from 0 to 10, with 10 being the worst. Patients are asked to categorize the result as excellent, very good, good, fair and poor.
Side effects and complications | 2 years postoperatively
  We will record any case of medical complications (embolism, cardiovascular event, pneumonia) and complications related to the surgical procedure (fractures, nerve injuries, deep and superficial infections, malpositioning of the components, instability, and dislocation) and revisions defined by removal or exchange of any component.
Cost-utility analysis | 2 years postoperatively
  In modern health economics, thresholds have been estimated for acceptable cost-utility ratios - the threshold for how much health care providers will pay for an extra quality- adjusted life year (QALY). In England and in Europe, the threshold for an extra QALY is set at 20,000-30,000 pounds and 30,000 Euros respectively. The cost utility of the Comprehensive Nano stemless shoulder arthroplasty will be compared with these thresholds and with the cost utility of the uncemented Comprehensive stemmed total shoulder arthroplasty. The EQ-5D will be used to estimate QALY for individual patients.
Length of hospital stay | 3 months postoperatively
  How long time the patients are hospitalized postoperatively. The data will be extracted from the medical records.
Discharge destination | 3 months postoperatively
  Whether the patients are discharged to home, rehabilitation or nursing home. The data will be extracted from the medical records.
Pain medication usage | 2 years postoperatively
  Which kind and how much pain medication each patients have used. The data will be extracted from the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Randall Kristensen Nyring, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Herlev and Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No
It is not the plan to make IPD available to other researchers.

REFERENCES:
- [Background] Andersen MR, Winther NS, Lind T, Schroder HM, Flivik G, Petersen MM. Low Preoperative BMD Is Related to High Migration of Tibia Components in Uncemented TKA-92 Patients in a Combined DEXA and RSA Study With 2-Year Follow-Up. J Arthroplasty. 2017 Jul;32(7):2141-2146. doi: 10.1016/j.arth.2017.02.032. Epub 2017 Feb 28. PMID 28410836
- [Background] Andersen MR, Winther N, Lind T, SchroDer H, Flivik G, Petersen MM. Monoblock versus modular polyethylene insert in uncemented total knee arthroplasty. Acta Orthop. 2016 Dec;87(6):607-614. doi: 10.1080/17453674.2016.1233654. Epub 2016 Sep 20. PMID 27649258
- [Background] Andersen MR, Winther NS, Lind T, Schroder HM, Mork Petersen M. Bone Remodeling of the Distal Femur After Uncemented Total Knee Arthroplasty-A 2-Year Prospective DXA Study. J Clin Densitom. 2018 Apr-Jun;21(2):236-243. doi: 10.1016/j.jocd.2017.05.001. Epub 2017 Sep 13. PMID 28918227
- [Background] Ban I, Troelsen A, Christiansen DH, Svendsen SW, Kristensen MT. Standardised test protocol (Constant Score) for evaluation of functionality in patients with shoulder disorders. Dan Med J. 2013 Apr;60(4):A4608. PMID 23651718
- [Background] Barvencik F, Gebauer M, Beil FT, Vettorazzi E, Mumme M, Rupprecht M, Pogoda P, Wegscheider K, Rueger JM, Pueschel K, Amling M. Age- and sex-related changes of humeral head microarchitecture: histomorphometric analysis of 60 human specimens. J Orthop Res. 2010 Jan;28(1):18-26. doi: 10.1002/jor.20957. PMID 19630001
- [Background] ten Broeke RH, Hendrickx RP, Leffers P, Jutten LM, Geesink RG. Randomised trial comparing bone remodelling around two uncemented stems using modified Gruen zones. Hip Int. 2012 Jan-Feb;22(1):41-9. doi: 10.5301/HIP.2012.9103. PMID 22383318
- [Background] Brolin TJ, Cox RM, Abboud JA, Namdari S. Stemless Shoulder Arthroplasty: Review of Early Clinical and Radiographic Results. JBJS Rev. 2017 Aug;5(8):e3. doi: 10.2106/JBJS.RVW.16.00096. No abstract available. PMID 28763354
- [Background] Bryant D, Litchfield R, Sandow M, Gartsman GM, Guyatt G, Kirkley A. A comparison of pain, strength, range of motion, and functional outcomes after hemiarthroplasty and total shoulder arthroplasty in patients with osteoarthritis of the shoulder. A systematic review and meta-analysis. J Bone Joint Surg Am. 2005 Sep;87(9):1947-56. doi: 10.2106/JBJS.D.02854. PMID 16140808
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327
- [Background] Dawson J, Fitzpatrick R, Carr A. Questionnaire on the perceptions of patients about shoulder surgery. J Bone Joint Surg Br. 1996 Jul;78(4):593-600. PMID 8682827
- [Background] Frich LH, Noergaard PM, Brorson S. Validation of the Danish version of Oxford Shoulder Score. Dan Med Bull. 2011 Nov;58(11):A4335. PMID 22047932
- [Background] Gartsman GM, Roddey TS, Hammerman SM. Shoulder arthroplasty with or without resurfacing of the glenoid in patients who have osteoarthritis. J Bone Joint Surg Am. 2000 Jan;82(1):26-34. doi: 10.2106/00004623-200001000-00004. PMID 10653081
- [Background] Gluer CC, Steiger P, Selvidge R, Elliesen-Kliefoth K, Hayashi C, Genant HK. Comparative assessment of dual-photon absorptiometry and dual-energy radiography. Radiology. 1990 Jan;174(1):223-8. doi: 10.1148/radiology.174.1.2294552.
- [Background] Guillemin F, Bombardier C, Beaton D. Cross-cultural adaptation of health-related quality of life measures: literature review and proposed guidelines. J Clin Epidemiol. 1993 Dec;46(12):1417-32. doi: 10.1016/0895-4356(93)90142-n. PMID 8263569
- [Background] Izquierdo R, Voloshin I, Edwards S, Freehill MQ, Stanwood W, Wiater JM, Watters WC 3rd, Goldberg MJ, Keith M, Turkelson CM, Wies JL, Anderson S, Boyer K, Raymond L, Sluka P; American Academy of Orthopedic Surgeons. Treatment of glenohumeral osteoarthritis. J Am Acad Orthop Surg. 2010 Jun;18(6):375-82. doi: 10.5435/00124635-201006000-00010. PMID 20511443
- [Background] Jensen CL, Petersen MM, Schroder HM, Flivik G, Lund B. Revision total knee arthroplasty with the use of trabecular metal cones: a randomized radiostereometric analysis with 2 years of follow-up. J Arthroplasty. 2012 Dec;27(10):1820-1826.e2. doi: 10.1016/j.arth.2012.04.036. Epub 2012 Jul 13. PMID 22795879
- [Background] Jensen CL, Petersen MM, Schroder HM, Lund B. Bone mineral density changes of the proximal tibia after revision total knee arthroplasty. A randomised study with the use of porous tantalum metaphyseal cones. Int Orthop. 2012 Sep;36(9):1857-63. doi: 10.1007/s00264-012-1601-y. Epub 2012 Jun 26. PMID 22733440
- [Background] Johnston PS, Creighton RA, Romeo AA. Humeral component revision arthroplasty: outcomes of a split osteotomy technique. J Shoulder Elbow Surg. 2012 Apr;21(4):502-6. doi: 10.1016/j.jse.2011.02.001. Epub 2011 May 19. PMID 21600792
- [Background] Kumar S, Sperling JW, Haidukewych GH, Cofield RH. Periprosthetic humeral fractures after shoulder arthroplasty. J Bone Joint Surg Am. 2004 Apr;86(4):680-9. doi: 10.2106/00004623-200404000-00003. PMID 15069130
- [Background] Karrholm J, Gill RH, Valstar ER. The history and future of radiostereometric analysis. Clin Orthop Relat Res. 2006 Jul;448:10-21. doi: 10.1097/01.blo.0000224001.95141.fe. PMID 16826090
- [Background] Karrholm J. Radiostereometric analysis of early implant migration - a valuable tool to ensure proper introduction of new implants. Acta Orthop. 2012 Dec;83(6):551-2. doi: 10.3109/17453674.2012.745352. Epub 2012 Nov 5. No abstract available. PMID 23126576
- [Background] Laursen MB, Nielsen PT, Soballe K. Bone remodelling around HA-coated acetabular cups : a DEXA study with a 3-year follow-up in a randomised trial. Int Orthop. 2007 Apr;31(2):199-204. doi: 10.1007/s00264-006-0148-1. Epub 2006 Jun 8. PMID 16761153
- [Background] Liew AS, Johnson JA, Patterson SD, King GJ, Chess DG. Effect of screw placement on fixation in the humeral head. J Shoulder Elbow Surg. 2000 Sep-Oct;9(5):423-6. doi: 10.1067/mse.2000.107089. PMID 11075327
- [Background] Lo IK, Litchfield RB, Griffin S, Faber K, Patterson SD, Kirkley A. Quality-of-life outcome following hemiarthroplasty or total shoulder arthroplasty in patients with osteoarthritis. A prospective, randomized trial. J Bone Joint Surg Am. 2005 Oct;87(10):2178-85. doi: 10.2106/JBJS.D.02198. PMID 16203880
- [Background] Lo IK, Griffin S, Kirkley A. The development of a disease-specific quality of life measurement tool for osteoarthritis of the shoulder: The Western Ontario Osteoarthritis of the Shoulder (WOOS) index. Osteoarthritis Cartilage. 2001 Nov;9(8):771-8. doi: 10.1053/joca.2001.0474. PMID 11795997
- [Background] Maloney WJ, Sychterz C, Bragdon C, McGovern T, Jasty M, Engh CA, Harris WH. The Otto Aufranc Award. Skeletal response to well fixed femoral components inserted with and without cement. Clin Orthop Relat Res. 1996 Dec;(333):15-26. PMID 8981879
- [Background] Marchetti ME, Houde JP, Steinberg GG, Crane GK, Goss TP, Baran DT. Humeral bone density losses after shoulder surgery and immobilization. J Shoulder Elbow Surg. 1996 Nov-Dec;5(6):471-6. doi: 10.1016/s1058-2746(96)80020-6. PMID 8981273
- [Background] Mazess RB, Barden HS. Measurement of bone by dual-photon absorptiometry (DPA) and dual-energy X-ray absorptiometry (DEXA). Ann Chir Gynaecol. 1988;77(5-6):197-203. PMID 3076046
- [Background] Mechlenburg I, Klebe TM, Dossing KV, Amstrup A, Soballe K, Stilling M. Evaluation of periprosthetic bone mineral density and postoperative migration of humeral head resurfacing implants: two-year results of a randomized controlled clinical trial. J Shoulder Elbow Surg. 2014 Oct;23(10):1427-36. doi: 10.1016/j.jse.2014.05.012. PMID 25220196
- [Background] Nelissen RG, Pijls BG, Karrholm J, Malchau H, Nieuwenhuijse MJ, Valstar ER. RSA and registries: the quest for phased introduction of new implants. J Bone Joint Surg Am. 2011 Dec 21;93 Suppl 3:62-5. doi: 10.2106/JBJS.K.00907. PMID 22262426
- [Background] Nuttall D, Haines JF, Trail IA. The early migration of a partially cemented fluted pegged glenoid component using radiostereometric analysis. J Shoulder Elbow Surg. 2012 Sep;21(9):1191-6. doi: 10.1016/j.jse.2011.07.028. Epub 2011 Nov 1. PMID 22047783
- [Background] Nuttall D, Birch A, Haines JF, Trail IA. Radiostereographic analysis of a shoulder surface replacement: does hydroxyapatite have a place? Bone Joint J. 2014 Aug;96-B(8):1077-81. doi: 10.1302/0301-620X.96B8.30534. PMID 25086124
- [Background] Nuttall D, Haines JF, Trail II. A study of the micromovement of pegged and keeled glenoid components compared using radiostereometric analysis. J Shoulder Elbow Surg. 2007 May-Jun;16(3 Suppl):S65-70. doi: 10.1016/j.jse.2006.01.015. Epub 2006 Aug 7. PMID 17493557
- [Background] Phipatanakul WP, Bowen JM, Jobe CM. Removal of well-fixed flanged humeral prostheses may require humeral expansion. J Shoulder Elbow Surg. 2009 Sep-Oct;18(5):724-7. doi: 10.1016/j.jse.2008.11.021. Epub 2009 Mar 21. PMID 19318282
- [Background] Rasmussen JV, Jakobsen J, Olsen BS, Brorson S. Translation and validation of the Western Ontario Osteoarthritis of the Shoulder (WOOS) index - the Danish version. Patient Relat Outcome Meas. 2013 Sep 18;4:49-54. doi: 10.2147/PROM.S50976. eCollection 2013. PMID 24133377
- [Background] Rasmussen JV, Olsen BS, Sorensen AK, Hrobjartsson A, Brorson S. Resurfacing hemiarthroplasty compared to stemmed hemiarthroplasty for glenohumeral osteoarthritis: a randomised clinical trial. Int Orthop. 2015 Feb;39(2):263-9. doi: 10.1007/s00264-014-2505-9. Epub 2014 Aug 27. PMID 25159010
- [Background] Rasmussen JV, Hole R, Metlie T, Brorson S, Aarimaa V, Demir Y, Salomonsson B, Jensen SL. Anatomical total shoulder arthroplasty used for glenohumeral osteoarthritis has higher survival rates than hemiarthroplasty: a Nordic registry-based study. Osteoarthritis Cartilage. 2018 May;26(5):659-665. doi: 10.1016/j.joca.2018.02.896. Epub 2018 Feb 21. PMID 29474992
- [Background] Rasmussen JV, Olsen BS, Al-Hamdani A, Brorson S. Outcome of Revision Shoulder Arthroplasty After Resurfacing Hemiarthroplasty in Patients with Glenohumeral Osteoarthritis. J Bone Joint Surg Am. 2016 Oct 5;98(19):1631-1637. doi: 10.2106/JBJS.15.00934. PMID 27707849
- [Background] Rasmussen JV, Polk A, Brorson S, Sorensen AK, Olsen BS. Patient-reported outcome and risk of revision after shoulder replacement for osteoarthritis. 1,209 cases from the Danish Shoulder Arthroplasty Registry, 2006-2010. Acta Orthop. 2014 Apr;85(2):117-22. doi: 10.3109/17453674.2014.893497. PMID 24650020
- [Background] Rasmussen JV, Polk A, Sorensen AK, Olsen BS, Brorson S. Outcome, revision rate and indication for revision following resurfacing hemiarthroplasty for osteoarthritis of the shoulder: 837 operations reported to the Danish Shoulder Arthroplasty Registry. Bone Joint J. 2014 Apr;96-B(4):519-25. doi: 10.1302/0301-620X.96B4.31850. PMID 24692621
- [Background] Ryd L, Albrektsson BE, Carlsson L, Dansgard F, Herberts P, Lindstrand A, Regner L, Toksvig-Larsen S. Roentgen stereophotogrammetric analysis as a predictor of mechanical loosening of knee prostheses. J Bone Joint Surg Br. 1995 May;77(3):377-83. PMID 7744919
- [Background] Sahota S, Sperling JW, Cofield RH. Humeral windows and longitudinal splits for component removal in revision shoulder arthroplasty. J Shoulder Elbow Surg. 2014 Oct;23(10):1485-91. doi: 10.1016/j.jse.2014.02.004. Epub 2014 Apr 22. PMID 24766791
- [Background] Singh JA, Sperling J, Buchbinder R, McMaken K. Surgery for shoulder osteoarthritis: a Cochrane systematic review. J Rheumatol. 2011 Apr;38(4):598-605. doi: 10.3899/jrheum.101008. Epub 2011 Jan 15. PMID 21239751
- [Background] Stilling M, Mechlenburg I, Amstrup A, Soballe K, Klebe T. Precision of novel radiological methods in relation to resurfacing humeral head implants: assessment by radiostereometric analysis, DXA, and geometrical analysis. Arch Orthop Trauma Surg. 2012 Nov;132(11):1521-30. doi: 10.1007/s00402-012-1580-x. Epub 2012 Jul 7. PMID 22773108
- [Background] Ten Brinke B, Beumer A, Koenraadt KLM, Eygendaal D, Kraan GA, Mathijssen NMC. The accuracy and precision of radiostereometric analysis in upper limb arthroplasty. Acta Orthop. 2017 Jun;88(3):320-325. doi: 10.1080/17453674.2017.1291872. Epub 2017 Mar 2. PMID 28464752
- [Background] Trozzi C, Kaptein BL, Garling EH, Shelyakova T, Russo A, Bragonzoni L, Martelli S. Precision assessment of model-based RSA for a total knee prosthesis in a biplanar set-up. Knee. 2008 Oct;15(5):396-402. doi: 10.1016/j.knee.2008.05.001. Epub 2008 Jul 16. PMID 18635360
- [Background] Valstar ER, Gill R, Ryd L, Flivik G, Borlin N, Karrholm J. Guidelines for standardization of radiostereometry (RSA) of implants. Acta Orthop. 2005 Aug;76(4):563-72. doi: 10.1080/17453670510041574. PMID 16195075
- [Background] Valstar E, Kaptein B, Nelissen R. Radiostereometry and new prostheses. Acta Orthop. 2012 Apr;83(2):103-4. doi: 10.3109/17453674.2012.678796. Epub 2012 Apr 11. No abstract available. PMID 22489889
- [Background] Van Thiel GS, Halloran JP, Twigg S, Romeo AA, Nicholson GP. The vertical humeral osteotomy for stem removal in revision shoulder arthroplasty: results and technique. J Shoulder Elbow Surg. 2011 Dec;20(8):1248-54. doi: 10.1016/j.jse.2010.12.013. Epub 2011 Mar 21. PMID 21420326
- [Background] Winther NS, Jensen CL, Jensen CM, Lind T, Schroder HM, Flivik G, Petersen MM. Comparison of a novel porous titanium construct (Regenerex(R)) to a well proven porous coated tibial surface in cementless total knee arthroplasty - A prospective randomized RSA study with two-year follow-up. Knee. 2016 Dec;23(6):1002-1011. doi: 10.1016/j.knee.2016.09.010. Epub 2016 Oct 19. PMID 27769563
- [Background] Winther N, Jensen C, Petersen M, Lind T, Schroder H, Petersen M. Changes in bone mineral density of the proximal tibia after uncemented total knee arthroplasty. A prospective randomized study. Int Orthop. 2016 Feb;40(2):285-94. doi: 10.1007/s00264-015-2852-1. Epub 2015 Jul 17. PMID 26183139
- [Derived] Nyring MRK, Olsen BS, Yilmaz M, Petersen MM, Flivik G, Rasmussen JV. Early migration of stemless and stemmed humeral components after total shoulder arthroplasty for osteoarthritis-study protocol for a randomized controlled trial. Trials. 2020 Oct 7;21(1):830. doi: 10.1186/s13063-020-04763-8. PMID 33028390